CLINICAL TRIAL: NCT03006926
Title: An Open-Label Phase 1b Trial of Lenvatinib Plus Pembrolizumab in Subjects With Hepatocellular Carcinoma
Brief Title: A Trial of Lenvatinib Plus Pembrolizumab in Participants With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-116; KEYNOTE 524 (Other: Merck); 2018-000522-55 (EudraCT Number)
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; E7080; lenvatinib; pembrolizumab; Japan
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- lenvatinib 8 or 12 mg plus pembrolizumab 200 mg (Experimental): Participants will receive oral lenvatinib at a starting dose of 8 or 12 milligrams (mg) once a day (QD) in combination with intravenous pembrolizumab 200 mg every 3 weeks (Q3W) on a 21-day treatment cycle. The starting dose of lenvatinib will be based on Baseline body weight. Participants weighing greater than or equal to 60 kilograms (kg) will receive 12 mg QD; participants weighing less than 60 kg will receive 8 mg QD.
  Interventions: Drug: lenvatinib; Drug: pembrolizumab (200 mg)

INTERVENTIONS:
Drug: lenvatinib — 4 mg capsules
Drug: pembrolizumab (200 mg) — 30-minute intravenous infusion

SUMMARY:
This is an open-label Phase 1b study designed to evaluate the tolerability and safety of lenvatinib in combination with pembrolizumab in participants with hepatocellular carcinoma (HCC). The study will evaluate objective response rate and duration of response by modified Response Evaluation Criteria In Solid Tumors (mRECIST) for HCC and Response Evaluation Criteria In Solid Tumors (RECIST 1.1) based on independent imaging review (IIR).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hepatocellular carcinoma (HCC)
* HCC for which no other appropriate therapy is available. Note: Expansion Part: No prior systemic therapy for advanced/unresectable HCC
* Stage B (not applicable for transarterial chemoembolization [TACE]), or stage C based on Barcelona Clinic Liver Cancer (BCLC) staging system
* At least 1 measurable target lesion according to modified Response Evaluation Criteria in Solid Tumors (mRECIST)
* Child-Pugh score A
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 1
* Total triiodothyronine (T3) or free T3 and free thyroxine (T4) are within normal limits. (control by thyroid replacement therapy is acceptable.) Participants with T3, free T3 or free T4 abnormalities at screening who are asymptomatic can be eligible
* Adequately controlled blood pressure
* Adequate renal function
* Adequate bone marrow function
* Adequate blood coagulation function
* Adequate liver function
* Males or females age ≥ 18 years at the time of informed consent
* Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol

Exclusion Criteria:

* Prior treatment with lenvatinib or any anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Active malignancy (except for HCC or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 36 months
* Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial
* Active infection (any infection requiring systemic treatment). Hepatitis B or C [HBV/HCV] is allowed
* Participants with CNS metastases are not eligible, unless they have completed local therapy (eg, whole brain radiation therapy [WBRT], surgery or radiosurgery) and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (eg, radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (6):
  - California Pacific Medical Center (CPMC), San Francisco, California
  - Ronald Reagan UCLA Medical Center, Santa Monica, California
  - Mercy Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine Mount Sinai, New York, New York
  - BRCR Global Texas, Edinburg, Texas
- France (4):
  - Hôpital Haut-Levêque Centre médico-chirurgical Magellan, Pessac, Bordeaux
  - Centre Eugène Marquis de Rennes, Rennes, Brittany Region
  - CHU Toulouse, Toulouse, Occitanie
  - Hôpital Timone, Marseille, Provence-Alpes-Côte d'Azur Region
- Italy (2):
  - IRCCS Istituto Clinico Humanitas, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna, Province of Bologna
- Japan (4):
  - Eisai Trial Site 2, Kashiwa, Chiba
  - Eisai Trial Site 4, Kawasaki, Kanagawa
  - Eisai Trial Site 3, Sayama, Osaka
  - Eisai Trial Site 1, Chuo-ku, Tokyo
- Russia (4):
  - Republican Clinical Oncology Dispensary, Ufa, Bashkortostan Republic
  - St. Petersburg City Clinical Oncology Dispansery, Saint Petersburg, Leningradskaya Oblast'
  - S.I. Russian Oncological Research Center n.a. N. N. Blokhin RAMS, Moscow, Moscow Oblast
  - Altay Regional Oncology Dispensary, Barnaul
- Spain (5):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Infanta Cristina de Badajoz, Badajoz, Province of Badajoz
  - Hospital Universitario de Salamanca, Salamanca, Province of Salamanca
- Royal Free Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finn RS, Ikeda M, Zhu AX, Sung MW, Baron AD, Kudo M, Okusaka T, Kobayashi M, Kumada H, Kaneko S, Pracht M, Mamontov K, Meyer T, Kubota T, Dutcus CE, Saito K, Siegel AB, Dubrovsky L, Mody K, Llovet JM. Phase Ib Study of Lenvatinib Plus Pembrolizumab in Patients With Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2020 Sep 10;38(26):2960-2970. doi: 10.1200/JCO.20.00808. Epub 2020 Jul 27. PMID 32716739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 24 investigative sites in the United States, Japan, United Kingdom, France, Italy, Spain, and Russian Federation from 13 February 2017 to 22 November 2022.
Pre-assignment Details: A total of 104 participants were enrolled and received treatment. Of these, 6 participants were enrolled in Dose Limiting Toxicity (DLT) part and 98 were enrolled in the expansion part.
Groups:
- DLT Part: Lenvatinib 12 mg or 8 mg + Pembrolizumab 200 mg: In the DLT part, participants received lenvatinib 12 milligram (mg) or 8 mg capsules, orally, once daily, in combination with pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in Cycle 1 of a 21-day treatment cycle. Participants with body weight greater than or equal to (>=) 60 kilogram (kg) received lenvatinib 12 mg; participants with body weight less than (<) 60 kg, received lenvatinib 8 mg. Participants who discontinued treatment in Cycle 1, entered the follow-up phase. Participants who were still receiving treatment at the end of Cycle 1, continued to receive same treatment until progressive disease (PD), development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor. Upon confirmation of the tolerability of the tested combination regimen of lenvatinib plus pembrolizumab in Cycle 1, expansion part was opened for participant's enrollment.
- Expansion Part: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg: In the Expansion part, participants received lenvatinib 12 mg or 8 mg capsules, orally, once daily, in combination with pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in 21-day treatment cycles until PD, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor. Participants with body weight >=60 kg received lenvatinib 12 mg; participants with body weight <60 kg, received lenvatinib 8 mg.
Period: Overall Study
Arm/Group | DLT Part: Lenvatinib 12 mg or 8 mg + Pembrolizumab 200 mg | Expansion Part: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Started | 6 | 98
Japanese Population | 6 | 16
Non-Japanese Population | 0 | 82
Completed | 6 | 0
Not Completed | 0 | 98
Not completed — Adverse Event | 0 | 27
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Radiological Disease Progression | 0 | 52
Not completed — Clinical Disease Progression | 0 | 10
Not completed — Other | 0 | 8

BASELINE CHARACTERISTICS:
Population: The efficacy analysis set included all participants who had received at least 1 dose of study drug.
Groups:
- DLT Part: Lenvatinib 12 mg or 8 mg + Pembrolizumab 200 mg: In the DLT part, participants received lenvatinib 12 mg or 8 mg capsules, orally, once daily, in combination with pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in Cycle 1 of a 21-day treatment cycle. Participants with body weight >=60 kg received lenvatinib 12 mg; participants with body weight <60 kg, received lenvatinib 8 mg. Participants who discontinued treatment in Cycle 1, entered the follow-up phase. Participants who were still receiving treatment at the end of Cycle 1, continued to receive same treatment until PD, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor. Upon confirmation of the tolerability of the tested combination regimen of lenvatinib plus pembrolizumab in Cycle 1, expansion part was opened for participant's enrollment.
- Total: Total of all reporting groups
Arm/Group | DLT Part: Lenvatinib 12 mg or 8 mg + Pembrolizumab 200 mg | Expansion Part: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 6 | 98 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.11) | 66.2 (8.16) | 66.1 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 19 | 20
  Male | 5 | 79 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 6 | 78 | 84
  Unknown or Not Reported | 0 | 17 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 26 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 0 | 51 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 19 | 19

OUTCOME MEASURES:

1. Primary Outcome: DLT Part: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an adverse event (AE) that emerged during the time from the first dose of study drug to 120 days (if participant initiated new anticancer therapy) following last dose of study drug, was absent at pretreatment (Baseline) or reemerged during treatment, was at pretreatment (Baseline) but stopped before treatment or worsened in severity during treatment relative to the pretreatment state, when AE was continuous. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening (that is, participant was at immediate risk of death from AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug).
Time Frame: From first dose until 120 days after the last dose (up to 50.2 months)
Population: The safety analysis set included all participants who had received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DLT Part: Lenvatinib 12 mg or 8 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Participants
  TEAEs | 6
  SAEs | 4

2. Primary Outcome: Expansion Part: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an AE that emerged during the time from the first dose of study drug to 120 days (if participant initiated new anticancer therapy) following last dose of study drug, was absent at pretreatment (Baseline) or reemerged during treatment, was at pretreatment (Baseline) but stopped before treatment or worsened in severity during treatment relative to the pretreatment state, when AE was continuous. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening (that is, participant was at immediate risk of death from AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug).
Time Frame: From first dose until 120 days after the last dose (up to 50.2 months)
Population: The safety analysis set included all participants who had received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Part: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 98
Participants
  TEAEs | 97
  SAEs | 73

3. Primary Outcome: DLT Part: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was graded according to Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03). DLT was defined as any of the following: (1) any of the hematological or nonhematological toxicities considered to be at least possibly related to lenvatinib and/or pembrolizumab occurring during Cycle 1; (2) failure to administer >=75 percent (%) of the planned dosage of lenvatinib as a result of treatment-related toxicity during Cycle 1; (3) participants who discontinued treatment due to treatment-related toxicity in Cycle 1; (4) greater than (>) 2 week delay in starting pembrolizumab in Cycle 2 because of a treatment-related toxicity, even if the toxicity did not meet DLT criteria.
Time Frame: From first dose of study drug up to Cycle 1 Day 21 (Cycle length= 21 days)
Population: The DLT analysis set included all participants (except for the Expansion part) who had completed Cycle 1 without major protocol deviation with at least 75% of study drug compliance and assessed for DLT, and participants who had experienced DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | DLT Part: Lenvatinib 12 mg or 8 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Participants | 0

4. Primary Outcome: DLT+Expansion Part: Objective Response Rate (ORR) Based on mRECIST and RECIST Version (v) 1.1 Assessed by Independent Imaging Review (IIR)
Description: ORR was defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) based on modified Response Evaluation Criteria in Solid Tumors (mRECIST) and Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 assessed by IIR analysis. Responses (PR or CR) were confirmed no less than 4 weeks after the initial response. CR defined as disappearance of all target lesions and non-target lesions (a short diameter is <10 millimeter [mm] if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the long diameter (LD) (hereafter referred to as sum of LD) of all target lesions, as compared with Baseline summed LD.
Time Frame: From the first dose of study drug to the first date of documentation of PD or death, whichever occurred first (up to 46.2 months)
Population: All participants with hepatocellular carcinoma (HCC) who had received at least 1 dose of combination of lenvatinib and pembrolizumab, as first line (1L) therapy, with no prior systemic therapy. In DLT part, 4 participants had received prior systemic therapy with sorafenib; therefore, they were excluded from analysis for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg: Participants received lenvatinib 8 or 12 mg, capsules, orally, once daily in combination with pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in 21-day treatment cycles as first line therapy until PD, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor. Participants with body weight >=60 kg received lenvatinib 12 mg; participants with body weight <60 kg, received lenvatinib 8 mg.
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 100
percentage of participants
  RECIST v1.1 | 38.0 [28.5 to 48.3]
  mRECIST | 46.0 [36.0 to 56.3]

5. Primary Outcome: DLT+Expansion Part: Duration of Response (DOR) Based on mRECIST Assessed by IIR
Description: DOR was defined as the time from the first documentation of CR or PR to the date of first documentation of PD or death (whichever occurred first) in participants with confirmed CR or PR based on mRECIST assessed by IIR analysis. CR defined as disappearance of all target lesions and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the LD (hereafter referred to as sum of LD) of all target and non-target lesions, as compared with Baseline summed LD. PD was defined as at least a 20% increase in the sum of LD of target and non-target lesions as compared with the smallest sum of LD, and the increase of LD was at least 5 mm (including new lesions).
Time Frame: From date of first documented confirmed CR or PR until date of first documentation of PD or death, whichever occurred first (up to 46.2 months)
Population: All participants with HCC who received at least 1 dose of combination of lenvatinib and pembrolizumab as 1L therapy with no prior systemic therapy. In DLT part, 4 participants who received prior systemic therapy with sorafenib were excluded from analysis for this measure. Overall number analyzed were the participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 46
months | 16.7 [8.6 to NA] — Upper limit of confidence interval could not be estimated due to an insufficient number of events.

6. Primary Outcome: DLT+Expansion Part: Duration of Response (DOR) Based on RECIST v1.1 Assessed by IIR
Description: DOR was defined as the time from the first documentation of CR or PR to the date of first documentation of PD or death (whichever occurred first) in participants with confirmed CR or PR based on RECIST v1.1 assessed by IIR analysis. CR defined as disappearance of all target lesions and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the LD (hereafter referred to as sum of LD) of all target and non-target lesions, as compared with Baseline summed LD. PD was defined as at least a 20% increase in the sum of LD of target and non-target lesions as compared with the smallest sum of LD, and the increase of LD was at least 5 mm (including new lesions).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 38
months | NA [12.6 to NA] — Median and upper limit of confidence interval could not be estimated due to an insufficient number of events.

7. Secondary Outcome: DLT+Expansion Part: Objective Response Rate (ORR) Based on mRECIST Assessed by Investigator Review
Description: ORR was defined as the percentage of participants who had BOR of CR or PR based on mRECIST assessed by investigator review. Responses (PR or CR) were confirmed no less than 4 weeks after the initial response. CR defined as disappearance of all target lesions and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the LD (hereafter referred to as sum of LD) of all target and non-target lesions, as compared with Baseline summed LD.
Time Frame: as for outcome 4
Population: All participants with HCC who had received at least 1 dose of combination of lenvatinib and pembrolizumab, as 1L therapy, with no prior systemic therapy. In DLT part of the study, 4 participants had received prior sorafenib; therefore, they were excluded from analysis for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HCC 1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg: Participants received lenvatinib 8 or 12 mg, capsules, orally, once daily in combination with pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in 21-day treatment cycles as first line therapy until PD, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor. Participants with body weight >=60 kg received lenvatinib 12 mg; participants with body weight <60 kg, received lenvatinib 8 mg.
Arm/Group | HCC 1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 100
percentage of participants | 43.0 [33.1 to 53.3]

8. Secondary Outcome: DLT+Expansion Part: Duration of Response (DOR) Based on mRECIST Assessed by Investigator Review
Description: DOR was defined as the time from the first documentation of CR or PR to the date of first documentation of PD or death (whichever occurred first) based on mRECIST assessed by investigator review. CR defined as disappearance of all target and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the LD (hereafter referred to as sum of LD) of all target and non-target lesions, as compared with Baseline summed LD. PD was defined as at least a 20% increase in the sum of LD of target and non-target lesions as compared with the smallest sum of LD, and the increase of LD was at least 5 mm (including new lesions).
Time Frame: as for outcome 5
Population: All participants with HCC who had received at least 1 dose of combination of lenvatinib and pembrolizumab, as 1L therapy, with no prior systemic therapy. In DLT part of study, 4 participants had received prior sorafenib; therefore, they were excluded. "Overall Number of Participants Analyzed": participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 43
months | 17.1 [6.9 to 19.3]

9. Secondary Outcome: DLT+Expansion Part: Progression-free Survival (PFS) Based on mRECIST and RECIST v1.1 Assessed by IIR and Based on mRECIST Assessed by Investigator Review
Description: PFS was defined as the time from the first study dose date to the date of first documentation of PD or death (whichever occurred first) based on mRECIST and RECIST v1.1 assessed by IIR, and mRECIST assessed by investigator review. PD was defined as at least a 20% increase in the sum of LD of target and non-target lesions as compared with the smallest sum of LD, and the increase of LD was at least 5 mm (including new lesions).
Time Frame: From the first study dose date to the date of first documentation of PD or death, whichever occurred first (up to 46.2 months)
Population: All participants with HCC who had received at least 1 dose of combination of lenvatinib and pembrolizumab, as 1L therapy, with no prior systemic therapy. In DLT part of the study, 4 participants had received prior systemic therapy with sorafenib; therefore, they were excluded from analysis for this measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 100
months
  mRECIST: IIR | 9.6 [5.6 to 11.8]
  RECIST v1.1: IIR | 9.6 [7.6 to 10.8]
  mRECIST: Investigator Review | 9.3 [7.4 to 9.8]

10. Secondary Outcome: DLT+Expansion Part: Time-to-Progression (TTP) Based on mRECIST and RECIST v1.1 Assessed by IIR and Based on mRECIST Assessed by Investigator Review
Description: TTP was defined as the time from the first study dose date to the date of first documentation of PD, based on mRECIST and RECIST v1.1 assessed by IIR and mRECIST assessed by an investigator review. PD was defined as at least a 20% increase in the sum of LD of target and non-target lesions as compared with the smallest sum of LD, and the increase of LD was at least 5 mm (including new lesions).
Time Frame: From date of first dose of study drug until PD (up to 46.2 months)
Population: All participants with HCC who had received at least 1 dose of combination of lenvatinib and pembrolizumab, as 1L therapy, with no prior systemic therapy. In DLT part of the study, 4 participants had received prior systemic therapy with sorafenib; therefore, they were excluded from analysis of this measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 100
months
  mRECIST: IIR | 9.9 [9.3 to 20.0]
  RECIST v1.1: IIR | 10.8 [9.6 to 24.3]
  mRECIST: Investigator Review | 9.8 [7.7 to 15.9]

11. Secondary Outcome: DLT+Expansion Part: Time-to-Response (TTR) Based on mRECIST Assessed by IIR
Description: TTR was defined as the time from the date of first study dose to the date of first documentation of CR or PR, in participants with confirmed CR or PR. It was evaluated according to mRECIST assessed by IIR. CR defined as disappearance of all target and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the LD (hereafter referred to as sum of LD) of all target and non-target lesions, as compared with Baseline summed LD.
Time Frame: From date of first dose of study drug until CR or PR (up to 46.2 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 46
months | 2.5 [1.2 to 7.6]

12. Secondary Outcome: DLT+Expansion Part: Time-to-Response (TTR) Based on RECIST v1.1 Assessed by IIR
Description: TTR was defined as the time from the date of first study dose to the date of first documentation of CR or PR, in participants with confirmed CR or PR. It was evaluated according to RECIST v1.1 assessed by IIR. CR defined as disappearance of all target and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the LD (hereafter referred to as sum of LD) of all target and non-target lesions, as compared with Baseline summed LD.
Time Frame: From date of first dose of study drug until CR or PR (up to 46.2 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 38
months | 2.8 [1.2 to 13.8]

13. Secondary Outcome: DLT+Expansion Part: Time-to-Response (TTR) Based on mRECIST Assessed by Investigator Review
Description: TTR was defined as the time from the date of first study dose to the date of first documentation of CR or PR, in participants with confirmed CR or PR. It was evaluated according to mRECIST assessed by investigator review. CR defined as disappearance of all target and non-target lesions (a short diameter is <10 mm if it exists in a lymph node). PR defined as at least 30% decrease in the sum of the LD (hereafter referred to as sum of LD) of all target and non-target lesions, as compared with Baseline summed LD.
Time Frame: From date of first dose of study drug until CR or PR (up to 46.2 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 43
months | 2.7 [1.2 to 15.7]

14. Secondary Outcome: DLT+Expansion Part: Overall Survival (OS)
Description: OS was measured from the date of first dose of study drug until date of death from any cause. Participants who were lost to follow-up or who were alive at the date of data cutoff were censored at the date the participants were last known alive, whichever came earlier.
Time Frame: From the date of first dose of study drug until date of death from any cause (up to 48.1 months)
Population: All participants with HCC who had received at least 1 dose of combination of lenvatinib and pembrolizumab, as 1L therapy, with no prior systemic therapy. In DLT part of study, 4 participants had received prior systemic therapy with sorafenib; therefore, they were excluded from analysis of this measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 100
months | 20.4 [14.4 to 25.9]

15. Secondary Outcome: DLT+Expansion Part, Cmax: Maximum Observed Plasma Concentration for Lenvatinib
Description: Cmax was defined as the maximum plasma concentration for lenvatinib. Cmax was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by liquid chromatography with tandem mass spectrometry (LC-MS/MS). As per pharmacokinetic (PK) planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=21 days)
Population: PK Analysis Set included all participants who had received at least 1 dose of lenvatinib and pembrolizumab and had evaluable concentration data (data within the limit of quantification). "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg: Japanese participants who received lenvatinib 8 mg capsules, orally, once daily in combination with pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in 21-day treatment cycles as first line therapy until PD, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
- DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg: Non-Japanese participants who received lenvatinib 8 mg capsules, orally, once daily in combination with pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in 21-day treatment cycles as first line therapy until PD, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
- DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg: Japanese participants who received lenvatinib 12 mg capsules, orally, once daily in combination with pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in 21-day treatment cycles as first line therapy until PD, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
- DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg: Non-Japanese participants who received lenvatinib 12 mg capsules, orally, once daily in combination with pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in 21-day treatment cycles as first line therapy until PD, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 7 | 1 | 11 | 9
nanogram per milliliter (ng/mL) | 127 (37.7) | 98.3 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 168 (29.7) | 145 (30.9)

16. Secondary Outcome: DLT+Expansion Part, Tmax: Time to Reach the Cmax for Lenvatinib
Description: Tmax was defined as the time to reach maximum observed plasma concentration (Cmax) for lenvatinib. Tmax was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 7 | 1 | 11 | 9
hours | 3.90 [1.00 to 7.97] | 4.00 [NA to NA] — Full Range (minimum and maximum) could not be calculated for a single participant. | 3.92 [0.82 to 7.92] | 4.00 [2.00 to 8.80]

17. Secondary Outcome: DLT+Expansion Part, AUC(0-t): Area Under the Plasma Concentration-time Curve From Zero Time to the Last Measurable Point for Lenvatinib
Description: AUC(0-t) was defined as the area under the plasma concentration-time curve from 0 time to last measurable point for lenvatinib. AUC(0-t) was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=21 days)
Population: PK Analysis Set included all participants who had received at least 1 dose of lenvatinib and pembrolizumab and had evaluable concentration data (data within the limit of quantification). "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure (with concentration data within the limit of quantification).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 7 | 0 | 11 | 4
nanogram*hour per milliliter (ng*h/mL) | 1230 (7.61) |  | 1690 (23.7) | 1950 (39.2)

18. Secondary Outcome: DLT+Expansion Part, AUC(0-ti): Area Under The Plasma Concentration-time Curve From Zero (Pre-Dose) to a Given Sampling Time (ti) for Lenvatinib
Description: AUC(0-ti) was defined as the area under the plasma concentration-time curve from 0 to a given sampling time for lenvatinib. AUC(0-ti) was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Days 1 and 15: 0-8 hours post-dose (Cycle length=21 days)
Population: PK Analysis Set included all participants who received at least 1 dose of lenvatinib and pembrolizumab and have evaluable concentration data (data within the limit of quantification). "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure (with concentration data within the limit of quantification) and "number analyzed" signifies participants who were evaluable for specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 7 | 0 | 11 | 6
ng*h/mL
  Cycle 1 Day 1: 0-8 hours post-dose | 673 (29.3) |  | 868 (25.9) | 736 (42.2)
  Cycle 1 Day 15: 0-8 hours post-dose: number analyzed (Participants) | 4 | 0 | 6 | 4
  Cycle 1 Day 15: 0-8 hours post-dose | 793 (36.0) |  | 1020 (57.4) | 1120 (18.2)

19. Secondary Outcome: DLT+Expansion Part, AUC(0-Inf): Area Under the Plasma Concentration-time Curve From Zero to Infinity for Lenvatinib
Description: AUC(0-Inf) was defined as the area under the plasma concentration-time curve from 0 to infinity for lenvatinib. AUC(0-Inf) was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Days 1 and 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 1 | 0 | 5 | 2
ng*h/mL
  Cycle 1 Day 1: 0-24 hours post-dose | 1340 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. |  | 1900 (31.8) | 1540 (16.6)
  Cycle 1 Day 15: 0-24 hours post-dose: number analyzed (Participants) | 0 | 0 | 1 | 1
  Cycle 1 Day 15: 0-24 hours post-dose |  |  | 4690 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 2530 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant.

20. Secondary Outcome: DLT+Expansion Part, t1/2: Terminal Elimination Phase Half-Life for Lenvatinib
Description: t1/2 was defined as the terminal elimination phase half-life for lenvatinib. t1/2 was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Days 1 and 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 1 | 0 | 5 | 2
hours
  Cycle 1 Day 1: 0-24 hours post-dose | 7.71 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. |  | 6.64 (16.0) | 5.75 (3.07)
  Cycle 1 Day 15: 0-24 hours post-dose: number analyzed (Participants) | 0 | 0 | 1 | 1
  Cycle 1 Day 15: 0-24 hours post-dose |  |  | 7.33 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 6.48 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant.

21. Secondary Outcome: DLT+Expansion Part, CL/F: Apparent Total Clearance for Lenvatinib
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F was calculated as (Dose/AUC(0-inf))/F. Where AUC(0-inf) is the area under the plasma concentration-time curve from zero to infinity and F is the bioavailability of the drug. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=21 days)
Population: PK Analysis Set included all participants who received at least 1 dose of lenvatinib and pembrolizumab and have evaluable concentration data (data within the limit of quantification). "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure (with concentration data within the limit of quantification).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 1 | 0 | 5 | 2
liter per hour (L/h) | 5.98 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. |  | 6.32 (31.6) | 7.79 (16.7)

22. Secondary Outcome: DLT+Expansion Part, Vz/F: Apparent Terminal Volume of Distribution for Lenvatinib
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F was calculated as (CL/F)/Lambda Z. Where, CL/F is the apparent total clearance and lambda Z is the apparent terminal elimination rate constant. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 1 | 0 | 5 | 2
liter | 66.6 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. |  | 60.6 (23.2) | 64.7 (19.8)

23. Secondary Outcome: DLT+Expansion Part, Css,Max: Maximum Observed Plasma Concentration at Steady State for Lenvatinib
Description: Css,max was defined as the maximum plasma concentration at steady state for lenvatinib. Css,max was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=21 days)
Population: PK Analysis Set included all participants who received at least 1 dose of lenvatinib and pembrolizumab and have evaluable concentration data (data within the limit of quantification). "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 4 | 1 | 8 | 5
ng/mL | 154 (25.1) | 145 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 201 (53.5) | 193 (17.8)

24. Secondary Outcome: DLT+Expansion Part, Css,Min: Minimum Observed Plasma Concentration at Steady State for Lenvatinib
Description: Css,min is the minimum plasma concentration at steady state for lenvatinib. Css,min was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 4 | 1 | 8 | 5
ng/mL | 42.9 (24.7) | 14.3 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 33.4 (48.1) | 34.3 (51.3)

25. Secondary Outcome: DLT+Expansion Part, Tss,Max: Time to Maximum Observed Concentration at Steady State For Lenvatinib
Description: Tss,Max was defined as the time to reach maximum observed plasma concentration of lenvatinib at steady state. Tss,Max was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 23
Measure: Median (Full Range); unit: hours
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 4 | 1 | 8 | 5
hours | 6.01 [4.00 to 8.00] | 4.02 [NA to NA] — Full Range (minimum and maximum) could not be calculated for a single participant. | 3.89 [2.02 to 7.77] | 4.00 [1.98 to 4.42]

26. Secondary Outcome: DLT+Expansion Part, AUC(0-tau): Area Under the Plasma Concentration-time Curve Over the Dosing Interval for Lenvatinib
Description: AUC(0-tau) was defined as the area under the plasma concentration-time curve over dosing interval for lenvatinib. AUC(0-tau) was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 0 | 0 | 1 | 3
ng*h/mL |  |  | 4150 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 2330 (16.5)

27. Secondary Outcome: DLT+Expansion Part, Clss/F: Apparent Total Clearance Following Oral Administration at Steady State for Lenvatinib
Description: Clearance of a drug at steady state is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CLss/F was calculated as (Dose/AUC(0-tau))/F. Where, AUC(0-tau) is the area under the plasma concentration-time curve over the dosing interval and F is the bioavailability of the drug. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 0 | 0 | 1 | 3
L/h |  |  | 2.89 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 5.14 (16.4)

28. Secondary Outcome: DLT+Expansion Part, Css,Av: Average Steady State Plasma Concentration for Lenvatinib
Description: Css,Av was defined as the average plasma concentration at steady state for lenvatinib. Css,Av was derived by non-compartmental analysis using lenvatinib plasma concentrations quantified by LC-MS/MS. Css,Av was calculated as AUC(0-tau)/tau. Where, AUC(0-tau) is the area under the plasma concentration-time curve over the dosing interval and tau is the length of dosing interval. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 0 | 0 | 1 | 3
ng/mL |  |  | 173 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 97.2 (16.4)

29. Secondary Outcome: DLT+Expansion Part, Vz,ss/F: Apparent Terminal Volume of Distribution at Steady State for Lenvatinib
Description: Volume of distribution at steady state was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz,ss/F was calculated as (CLss/F)/Lambda Z. Where, CLss/F is the apparent total clearance following oral administration at steady state and lambda Z is the apparent terminal elimination rate constant. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 0 | 0 | 1 | 1
liter |  |  | 30.6 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 48.5 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant.

30. Secondary Outcome: DLT+Expansion Part, Rac (Cmax): Accumulation Ratio of Cmax for Lenvatinib
Description: Rac(Cmax) was calculated as Css,max at Cycle 1 Day 15/Cmax at Cycle 1 Day 1. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Days 1 and 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 4 | 1 | 8 | 5
ratio | 1.07 (28.6) | 1.48 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 1.17 (33.9) | 1.38 (41.7)

31. Secondary Outcome: DLT+Expansion Part, Rac (AUC0-8 Hour): Accumulation Ratio of AUC(0-8 Hour) for Lenvatinib
Description: Rac(AUC0-8 hour) was calculated as AUC(0-8 hour) at Cycle 1 Day 15/AUC(0-8 hour) at Cycle 1 Day 1. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Days 1 and 15: 0-8 hours post-dose (Cycle length=21 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 4 | 0 | 6 | 3
ratio | 1.07 (21.2) |  | 1.32 (44.8) | 1.83 (66.8)

32. Secondary Outcome: DLT+Expansion Part, %PTF: Percent (%) Peak-trough Fluctuation for Lenvatinib
Description: The PTF within complete dosing interval at steady state, calculated as PTF (%) = ([Css,max - Css,min]/Css,Av)* 100. Where, Css,max is the maximum observed plasma concentration at steady state and Css,min is the minimum observed plasma concentration at steady state and Css,Av average steady state plasma concentration. As per PK planned analysis for lenvatinib and as per sponsor's practice, the lenvatinib PK data was collected, analyzed and summarized according to Japanese and non-Japanese population in this study.
Time Frame: Cycle 1 Day 15: 0-24 hours post-dose (Cycle length=21 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage fluctuation
Arm/Group | DLT+Expansion Part, Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 8 mg | DLT+Expansion Part, Japanese Participants: Lenvatinib 12 mg | DLT+Expansion Part, Non-Japanese Participants: Lenvatinib 12 mg
Number analyzed (Participants) | 0 | 0 | 1 | 3
percentage fluctuation |  |  | 161 (NA) — Geometric Coefficient of Variation could not be calculated for a single participant. | 161 (34.0)

33. Secondary Outcome: DLT+Expansion Part, Ctrough: Trough (Pre-dose) Serum Concentration for Pembrolizumab
Description: Ctrough was defined as trough (pre-dose) serum concentration for pembrolizumab at steady state.
Time Frame: Cycles 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36: Pre-dose (each Cycle length=21 days)
Population: PK Analysis Set included all participants who had received at least 1 dose of pembrolizumab and had evaluable concentration data. "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for specified timepoints. As per PK planned analysis for pembrolizumab, the combined PK data for pembrolizumab was collected and analyzed for participants of DLT and Expansion part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Groups:
- DLT+Expansion Part: Pembrolizumab 200 mg: Participants received pembrolizumab 200 mg, infusion, intravenously, every 3 weeks, in 21-day treatment cycles as first line therapy until PD, development of unacceptable toxicity, withdrawal of consent, or study termination by sponsor.
Arm/Group | DLT+Expansion Part: Pembrolizumab 200 mg
Number analyzed (Participants) | 101
microgram per milliliter (mcg/mL)
  Cycle 1: Pre-dose | 0.00 (0.00)
  Cycle 2: Pre-dose: number analyzed (Participants) | 93
  Cycle 2: Pre-dose | 12.3 (40.7)
  Cycle 4: Pre-dose: number analyzed (Participants) | 76
  Cycle 4: Pre-dose | 21.9 (56.6)
  Cycle 6: Pre-dose: number analyzed (Participants) | 75
  Cycle 6: Pre-dose | 25.0 (64.7)
  Cycle 8: Pre-dose: number analyzed (Participants) | 59
  Cycle 8: Pre-dose | 26.6 (86.1)
  Cycle 12: Pre-dose: number analyzed (Participants) | 53
  Cycle 12: Pre-dose | 27.9 (57.7)
  Cycle 16: Pre-dose: number analyzed (Participants) | 37
  Cycle 16: Pre-dose | 33.6 (39.3)
  Cycle 20: Pre-dose: number analyzed (Participants) | 35
  Cycle 20: Pre-dose | 27.9 (50.1)
  Cycle 24: Pre-dose: number analyzed (Participants) | 27
  Cycle 24: Pre-dose | 29.0 (69.9)
  Cycle 28: Pre-dose: number analyzed (Participants) | 18
  Cycle 28: Pre-dose | 32.4 (49)
  Cycle 32: Pre-dose: number analyzed (Participants) | 7
  Cycle 32: Pre-dose | 30.7 (34.3)
  Cycle 36: Pre-dose: number analyzed (Participants) | 8
  Cycle 36: Pre-dose | 34.6 (40.2)

34. Secondary Outcome: DLT+Expansion Part: Number of Participants Positive for Serum Anti-drug Antibodies (ADA) Status
Description: ADA positive was defined as participants with at least one pre-treatment or post-dose sample positive in the confirmatory assay for antibodies against pembrolizumab. ADA was assessed using a validated electrochemiluminescence (ECL) immunoassay.
Time Frame: Cycles 1 and 6 Day 1: Pre-dose (each cycle length=21 days)
Population: All participants with HCC who received at least 1 dose of combination of lenvatinib and pembrolizumab as 1L therapy with no prior systemic therapy. Here, "overall number of participants analyzed" signifies participants with at least one ADA sample available after treatment with pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | HCC-1L: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
Number analyzed (Participants) | 81
Participants
  Cycle 1 Day 1: Pre-dose | 3
  Cycle 6 Day 1: Pre-dose | 0

ADVERSE EVENTS:
Time Frame: From the date of administration of the first dose of the study drug up to 120 days after the last dose of study drug (up to 50.2 months)
Description: The safety analysis set included all participants who had received at least 1 dose of study drug.
Arm/Group | DLT Part: Lenvatinib 12 mg or 8 mg + Pembrolizumab 200 mg | Expansion Part: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 5/6 | 67/98
Serious Adverse Events (participants affected / at risk) | 4/6 | 73/98
Other Adverse Events (participants affected / at risk) | 6/6 | 97/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLT Part: Lenvatinib 12 mg or 8 mg + Pembrolizumab 200 mg (N=6) | Expansion Part: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg (N=98)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 5 (6)
Death (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 2 (3)
Asthenia (General disorders) | 0 (0) | 2 (3)
Fatigue (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 3 (4)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (3)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 2 (2)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 4 (5)
Sepsis (Infections and infestations) | 0 (0) | 2 (3)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (3)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 9 (18)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (6)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 6 (11)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (3)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (3)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (3)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Dementia with Lewy bodies (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLT Part: Lenvatinib 12 mg or 8 mg + Pembrolizumab 200 mg (N=6) | Expansion Part: Lenvatinib 12 mg or 8 mg+ Pembrolizumab 200 mg (N=98)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 28 (79)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 10 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 13 (26)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 7 (7)
Hypothyroidism (Endocrine disorders) | 4 (4) | 31 (39)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 20 (30)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 10 (16)
Ascites (Gastrointestinal disorders) | 0 (0) | 12 (15)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 15 (19)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (15) | 58 (132)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 7 (7)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 20 (34)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 16 (27)
Vomiting (Gastrointestinal disorders) | 2 (3) | 18 (30)
Asthenia (General disorders) | 0 (0) | 27 (55)
Fatigue (General disorders) | 2 (2) | 37 (75)
Malaise (General disorders) | 1 (1) | 6 (17)
Oedema peripheral (General disorders) | 3 (4) | 20 (27)
Pyrexia (General disorders) | 0 (0) | 11 (18)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 10 (27)
Contrast media allergy (Immune system disorders) | 1 (1) | 1 (1)
Contrast media reaction (Immune system disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 9 (12)
Paronychia (Infections and infestations) | 1 (1) | 2 (2)
Rash pustular (Infections and infestations) | 0 (0) | 5 (8)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 6 (8)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 3 (5)
Alanine aminotransferase increased (Investigations) | 2 (5) | 21 (46)
Amylase increased (Investigations) | 0 (0) | 15 (44)
Aspartate aminotransferase increased (Investigations) | 2 (9) | 32 (103)
Blood albumin decreased (Investigations) | 0 (0) | 5 (6)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 16 (32)
Blood bilirubin increased (Investigations) | 0 (0) | 20 (77)
Blood creatinine increased (Investigations) | 0 (0) | 15 (38)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 6 (9)
Blood pressure increased (Investigations) | 0 (0) | 5 (8)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (2) | 8 (12)
Blood urea increased (Investigations) | 0 (0) | 6 (11)
C-reactive protein increased (Investigations) | 1 (1) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 9 (14)
Eosinophil count increased (Investigations) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 10 (22)
Lipase increased (Investigations) | 0 (0) | 23 (62)
Neutrophil count decreased (Investigations) | 3 (17) | 8 (54)
Platelet count decreased (Investigations) | 1 (3) | 13 (54)
Weight decreased (Investigations) | 4 (14) | 33 (76)
White blood cell count decreased (Investigations) | 1 (6) | 9 (60)
Decreased appetite (Metabolism and nutrition disorders) | 6 (16) | 37 (73)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 6 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 21 (67)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 8 (20)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 10 (29)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 19 (65)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 19 (30)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (7) | 20 (29)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 12 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 19 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (16)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 10 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 7 (13)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 9 (10)
Headache (Nervous system disorders) | 0 (0) | 10 (10)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 6 (10)
Insomnia (Psychiatric disorders) | 2 (2) | 8 (9)
Haematuria (Renal and urinary disorders) | 0 (0) | 8 (14)
Proteinuria (Renal and urinary disorders) | 2 (16) | 29 (79)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 10 (12)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 22 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (18)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 23 (48)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 22 (26)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 15 (23)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (19) | 46 (114)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 7 (11)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 5 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 5 (7)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (3) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 5 (12)
Lymphocyte count decreased (Investigations) | 0 (0) | 5 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 8 (14)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Renal impairment (Renal and urinary disorders) | 1 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT03006926/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03006926/SAP_001.pdf